CLINICAL TRIAL: NCT05203302
Title: Novel Coding Strategies for Children With Cochlear Implants
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 18-00437
Record Dates: First submitted 2022-01-10; First posted 2022-01-24 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-04

CONDITIONS: Deafness
MeSH Terms: conditions — Deafness

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Late Adult Cochlear Implant (LateAdultCI) (Experimental): Post-lingually implanted adults, 18+ years
  Interventions: Other: Single-Electrode Pulse Train; Other: Modulation Detection Threshold (MDT) and Gap Detection Tasks; Other: Sound coding strategy.
- Early Child Cochlear Implant (EarlyChildCI) (Experimental): Early implanted children, ages 7-17 years
  Interventions: Other: Modulation Detection Threshold (MDT) and Gap Detection Tasks; Other: Sound coding strategy.; Other: Electric-only spectral resolution
- Early Adult Cochlear Implant (EarlyAdultCI) (Experimental): Early implanted adults, ages 18 to 35 years
  Interventions: Other: Single-Electrode Pulse Train; Other: Sound coding strategy.
- Cochlear Implant (CI) (Experimental): CI children, ages 7-17 years, with aided residual hearing (bimodal/contralateral, electric+acoustic/ipsilateral)
  Interventions: Other: Electric-only spectral resolution
- Normal Hearing Children (NHC) (Active Comparator): Ages 7-17 years, Control Group
  Interventions: Other: Modulation Detection Threshold (MDT) and Gap Detection Tasks
- Normal Hearing Adults (NHA) (Active Comparator): 18+ years, Control Group
  Interventions: Other: Modulation Detection Threshold (MDT) and Gap Detection Tasks

INTERVENTIONS:
Other: Single-Electrode Pulse Train — AIM 2 - Stimuli will be presented on one of three electrodes (apical, middle, and basal) at an amplitude between 10 and 100% dynamic range in µAs in 10% dynamic range steps. Stimulation will be delivered at a rate of 1000 pps. The process will be repeated in random order until 20 loudness estimates are obtained for each stimulus (3 electrodes x 2 rates x 10 amplitudes) for each subject. The dynamic range will be determined by measuring the maximum acceptable loudness (MAL) and threshold for each of the stimuli. MAL will be measured by slowly raising the current level for each stimulus until the subject reports that it is as loud as they are willing to accept without becoming uncomfortably loud.
  Arms: Early Adult Cochlear Implant (EarlyAdultCI); Late Adult Cochlear Implant (LateAdultCI)
Other: Modulation Detection Threshold (MDT) and Gap Detection Tasks — AIM 1 - MDT will be set at 150 Hz. Testing will be conducted in soundfield in a sound booth at 60 dB Sound Pressure Level (SPL) while the participant listens with both implants adjusted to user setting.
  Arms: Early Child Cochlear Implant (EarlyChildCI); Late Adult Cochlear Implant (LateAdultCI); Normal Hearing Adults (NHA); Normal Hearing Children (NHC)
Other: Sound coding strategy. — Aim3 - Spectral-temporally modulated ripple test (SMRT), Quick Spectral Modulation Detection (QSMD), Modulation Detection, Gap Detection. CNC words will be set in quiet and Az-Bio/BabyBio sentences in quiet and multi-talker babble (+10 and +5 dB SNR) using both the subject's clinical map and the new reduced channels map. Tests will be presented in the soundfield at 60 dB SPL
  Arms: Early Adult Cochlear Implant (EarlyAdultCI); Early Child Cochlear Implant (EarlyChildCI); Late Adult Cochlear Implant (LateAdultCI)
Other: Electric-only spectral resolution — Aim 1- Spectral resolution will be tested using frequency allocations consisting of the full default clinical range as well as the subject's clinical frequency allocation if they differ. For Hybrid electrode users in which electrode contacts are closer in proximity in the cochlea, maps with a frequency allocation of 938-7938 Hz will also be tested in that it will closely approximate the frequency spacing of a Nucleus Contour Advance electrode array. Spectral resolution will be measured with three repetitions of the SMRT and one repetition of the QSMD test. Testing will be presented at 60 dB SPL in the soundfield with the acoustic ear plugged and muffed.
  Arms: Cochlear Implant (CI); Early Child Cochlear Implant (EarlyChildCI)

SUMMARY:
The purpose of this study is to understand performance with a cochlear implant. The long-term goals of this research are to improve sound perception with cochlear implants and to better understand the functioning of the auditory system. Information from individuals with and without cochlear implants will be compared.

DETAILED DESCRIPTION:
The overall objectives of this research are to 1) gain a better understanding of fundamental psychophysical abilities with electrical stimulation as a function of age (child vs adult), age at onset of deafness (pre- vs post-lingual), and acoustic hearing (normal vs limited or residual); and 2) determine whether manipulations in CI coding strategies will improve psychophysical and speech recognition outcomes for early implanted children. This work is expected to provide new insights into the corresponding improvements in perceptual outcomes to these newer strategies have been modest at best and performance has begun to level off.

ELIGIBILITY:
Inclusion Criteria:

* Be 7 years of age or older and pre-lingually implanted with a cochlear implant (before the age of 2 years), have aided residual hearing, or have normal hearing.
* Be ages 18 or older and post-lingually implanted or have normal hearing.
* Be ages 18-35 and pre-lingually implanted.

Exclusion Criteria:

* Any child implanted post-lingually

Ages: 6 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 190 (Estimated)
Dates: Start 2018-07-12 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Change in loudness growth in Cochlear Implant participants | Baseline Visit (Day 1) , Visit week 10
  Power functions will be fit for each of the loudness growth curves. Data will be analyzed using a mixed-design ANOVA with the two groups as the between-subjects factor and electrode and rate as within-subject factors.
Change in temporal resolution in Cochlear implant participants | Baseline Visit (Day 1) , Visit week 10
  A mixed-effect ANOVA will be conducted to determine if there is an effect of age group (children vs adults) and hearing condition (CI vs NH) for both modulation detection and gap detection tasks. Post-hoc two-sample t-tests will compare differences between NH and CI children as well as NH and CI adults. Post-hoc paired t-tests will compare differences between adults and children for both the NH and the CI populations.
Change in spectral resolution in Cochlear implant participants | Baseline Visit (Day 1) , Visit week 10
  A one-way ANOVA will be used to calculate the differences between the four groups. If significant, post-hoc t-tests will be performed using Rom's modified Bonferroni Type I error correction.
Difference in performance between the reduced channel map and the full map | Baseline Visit (Day 1) , Visit week 10
  A mixed-design ANOVA will be conducted for each of the tests with subject population as the between-subjects factor and sound coding strategy as the within-subjects factor

CONTACTS AND LOCATIONS:
Overall Officials: David M Landsberger, MD, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research. The investigator who proposed to use the data. The investigator who proposed to use the data.
Access Criteria: Upon reasonable request.Requests should be directed to natalia.stupak@nyulangone.org. To gain access, data requestors will need to sign a data access agreement.